CLINICAL TRIAL: NCT06295510
Title: A Cross-sectional Observational Study of the Association Between Food Intake and Endometrial Polyps
Brief Title: Observational Study of the Association Between Food Intake and Endometrial Polyps
Status: Not yet recruiting | Type: Observational
Sponsor: qinxiu zhang (Other)
Responsible Party: Sponsor-Investigator, qinxiu zhang, Head of ENT, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Other Study IDs: CDUTCM20240223
Record Dates: First submitted 2024-02-22; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Diet Habit; Endometrial Polyp; Women
Keywords: Diet; Endometrial polyp; Women; Milk tea
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy group (HG): Participants were grouped according to their basic conditions without any intervention.
  no intervention It's only observational study. No interventions.
  Interventions: Other: No interventions.
- case group（PG）: Participants were grouped according to their basic conditions without any intervention.
  no intervention It's only observational study. No interventions.
  Interventions: Other: No interventions.

INTERVENTIONS:
Other: No interventions. — It's only observational study.

SUMMARY:
There are currently no studies evaluating the association between diet and the incidence of endometrial polyps. We aim to evaluate the association to provide more recommendations for the early prevention of endometrial polyps.

DETAILED DESCRIPTION:
The incidence of endometrial polyps is closely related to daily diet and living habits. Due to the excessive use of food additives, the content of some common dietary hormones exceeds the standard, causing irreversible effects on female growth and development.

The daily diet structure is closely related to women's health, and the enrichment of estrogen in common drinks may cause adverse effects such as premature puberty in women, abnormal thyroid function, and changes in uterine structure. Therefore, the researchers conducted a retrospective analysis of patients with endometrial polyps and normal women to compare the associations and differences between daily diet and disease.

ELIGIBILITY:
Inclusion Criteria:

* Consistent with the international clinical diagnosis of endometrial polyps.Can complete content recall alone.

Exclusion Criteria:

* No other mental diseases. Not associated with other major diseases, including tumors, immune system diseases

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study period will include all patients who attended gynecological outpatient clinics between March 1, 2024 and May 1, 2024
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Hormonal dietary intake | Within the past 1 year
  Daily dietary intake questionnaire was used to evaluate.Weekly intake of milk tea, coffee, beverage, etc
Comparison of daily living habits | Within the past 1 year
  Sleep, exercise, and other basic information were assessed based on a daily habits questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Qinxiu Zhang, Study Director — Chengdu University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No
Readers can access the survey data through a public data platform

REFERENCES:
- [Derived] Fu R, Zhang S, Cai C, Wang X, Jiang Y, Zhuang X, Zhang J, Ji X, Yang C. Association between the intake of potentially risky beverages and the occurrence of endometrial polyps: a case-control study. Front Nutr. 2025 Feb 4;12:1538405. doi: 10.3389/fnut.2025.1538405. eCollection 2025. PMID 39968393